CLINICAL TRIAL: NCT07380425
Title: Effects of Pressure Support and Positive End-Expiratory Pressure Added to Deep Breathing Preoxygenation on Gastric Distension in Obese Patients: A Randomized Controlled Trial
Brief Title: Deep Breathing With and Without Pressure Support and PEEP for Preoxygenation in Obese Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Cagin Tanriverdi, Principal Investigator, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PamukkaleUCTanriverdi-002
Record Dates: First submitted 2026-01-11; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Obesity
Keywords: Preoxygenation; obesity; Pressure Support Ventilation; Positive End-Expiratory Pressure; Gastric Antrum Area
MeSH Terms: conditions — Obesity | interventions — Positive-Pressure Respiration

STUDY DESIGN:
Intervention Model Description: Three-arm parallel-group randomized trial comparing deep breathing alone, deep breathing with pressure support, and deep breathing with pressure support plus PEEP for preoxygenation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DB (Deep Breathing) (Experimental): Deep breathing preoxygenation with 100% oxygen at 12 L/min using.
  Interventions: Procedure: Positive End-Expiratory Pressure
- DB+PSV (Experimental): Preoxygenation with deep breathing supported by pressure-supported ventilation (PSV-Pro) with 12 cmH₂O pressure support and 100% oxygen at 12 L/min until EtO₂ reached 90%.
  Interventions: Procedure: Deep Breathing Preoxygenation
- DB+PSV+PEEP (Experimental): Deep breathing preoxygenation supported by PSV-Pro (pressure support 12 cmH₂O) with the addition of PEEP 6 cmH₂O; 100% oxygen at 12 L/min. This arm differs from Arm 2 by the application of PEEP.
  Interventions: Procedure: Pressure Support Ventilation

INTERVENTIONS:
Procedure: Deep Breathing Preoxygenation — Preoxygenation performed with deep breathing using a ventilator delivering 100% oxygen at a flow rate of 12 L/min.
  Arms: DB+PSV
Procedure: Pressure Support Ventilation — Application of pressure support ventilation with a pressure support level of 12 cmH₂O during preoxygenation.
  Arms: DB+PSV+PEEP
Procedure: Positive End-Expiratory Pressure — Application of positive end-expiratory pressure at a level of 6 cmH₂O during preoxygenation.
  Arms: DB (Deep Breathing)

SUMMARY:
Obese patients are at increased risk of low oxygen levels during the induction of general anesthesia. Preoxygenation with a face mask before anesthesia is routinely used to increase oxygen reserves. This study compares three preoxygenation techniques: deep breathing alone, deep breathing with pressure-supported ventilation, and deep breathing with pressure-supported ventilation plus positive end-expiratory pressure (PEEP).

The main goal of the study is to determine how quickly each technique allows patients to reach an adequate level of oxygen in the lungs. In addition, the study evaluates whether these techniques cause gastric distension, which could increase the risk of regurgitation. Gastric ultrasound is used to assess stomach size before and after preoxygenation.

The results of this study will help identify the most effective and safest method of preoxygenation in obese patients undergoing elective surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Obesity
* Scheduled for elective surgery under general anesthesia
* Able to cooperate with deep breathing during preoxygenation

Exclusion Criteria:

* Hemodynamic instability
* Poor cooperation
* Preoperative oxygen therapy requirement
* Conditions in which positive pressure ventilation may be harmful (e.g., increased intracranial or intraocular pressure)
* Pregnancy
* Emergency surgery
* Beard (preventing adequate face mask seal)
* Previous gastric surgery
* Inability to visualize the gastric antrum by ultrasonography

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-07-25 (Actual); Study Completion 2022-07-25 (Actual)

PRIMARY OUTCOMES:
Time to reach an end-tidal oxygen concentration (EtO₂) of 90% | Periprocedural (during the preoxygenation period, prior to induction of anesthesia)
  The time, in seconds, from the start of preoxygenation until the end-tidal oxygen concentration (EtO₂) reached 90%. End-tidal oxygen was measured at 30-second intervals using the anesthesia machine gas analyzer. Reaching EtO₂ 90% was defined as the endpoint of the preoxygenation period.

SECONDARY OUTCOMES:
Heart rate | Periprocedural (baseline and pre-induction)
  Heart rate was measured at baseline (before the start of preoxygenation) and at the end of the preoxygenation period, defined as the time point when end-tidal oxygen concentration (EtO₂) reached 90%.
Gastric antral cross-sectional area | Periprocedural (baseline and pre-induction)
  Gastric antral cross-sectional area measured by ultrasonography using a 2-5 MHz convex probe, calculated as (anteroposterior diameter × craniocaudal diameter × π)/4. Measurements were performed at baseline (before the start of preoxygenation) and at the completion of the preoxygenation period, defined as the time point when end-tidal oxygen concentration (EtO₂) reached 90%.
Gastric distension score | Periprocedural (baseline and pre-induction)
  Epigastric gastric distension assessed using a 4-point ordinal scale (0 = none, 1 = mild, 2 = moderate, 3 = marked). The score was recorded at baseline (before the start of preoxygenation) and at the completion of the preoxygenation period, defined as the time point when end-tidal oxygen concentration (EtO₂) reached 90%.
Reflux, belching, and discomfort | Periprocedural (baseline and pre-induction)
  Patient-reported occurrence of discomfort, symptomatic gastroesophageal reflux, or belching during the preoxygenation period. Events were assessed and recorded at the completion of the preoxygenation period, defined as the time point when end-tidal oxygen concentration (EtO₂) reached 90%.
Systolic Blood Pressure | Periprocedural (baseline and pre-induction)
  Systolic blood pressure measured noninvasively at baseline (before the start of preoxygenation) and at the completion of the preoxygenation period, defined as the time point when end-tidal oxygen concentration (EtO₂) reached 90%.
Diastolic Blood Pressure | Pre-induction (baseline and at completion of preoxygenation, defined by EtO₂ reaching 90%)
  Diastolic blood pressure measured noninvasively at baseline (before the start of preoxygenation) and at the completion of the preoxygenation period, defined as the time point when end-tidal oxygen concentration (EtO₂) reached 90%.
Peripheral Oxygen Saturation (SpO₂) | Periprocedural (baseline and pre-induction)
  Peripheral oxygen saturation (SpO₂) measured at baseline (before the start of preoxygenation) and at the completion of the preoxygenation period, defined as the time point when end-tidal oxygen concentration (EtO₂) reached 90%.

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Abou-Arab O, Guinot PG, Dimov E, Diouf M, de Broca B, Biet A, Zaatar R, Bernard E, Dupont H, Lorne E. Low-positive pressure ventilation improves non-hypoxaemic apnoea tolerance during ear, nose and throat pan-endoscopy: A randomised controlled trial. Eur J Anaesthesiol. 2016 Apr;33(4):269-74. doi: 10.1097/EJA.0000000000000394. PMID 26716862
- [Result] Taxak S, Gupta M, Bala R, Govil V, Lallar A. A prospective randomized study to evaluate the efficacy of pressure support ventilation with and without positive end expiratory pressure for preoxygenation in adult patients. Med Gas Res. 2023 Oct-Dec;13(4):187-191. doi: 10.4103/2045-9912.372665. PMID 37077116
- [Result] Hanouz JL, Lammens S, Tasle M, Lesage A, Gerard JL, Plaud B. Preoxygenation by spontaneous breathing or noninvasive positive pressure ventilation with and without positive end-expiratory pressure: A randomised controlled trial. Eur J Anaesthesiol. 2015 Dec;32(12):881-7. doi: 10.1097/EJA.0000000000000297. PMID 26225498
- [Result] Delay JM, Sebbane M, Jung B, Nocca D, Verzilli D, Pouzeratte Y, Kamel ME, Fabre JM, Eledjam JJ, Jaber S. The effectiveness of noninvasive positive pressure ventilation to enhance preoxygenation in morbidly obese patients: a randomized controlled study. Anesth Analg. 2008 Nov;107(5):1707-13. doi: 10.1213/ane.0b013e318183909b. PMID 18931236
- [Result] Nimmagadda U, Chiravuri SD, Salem MR, Joseph NJ, Wafai Y, Crystal GJ, El-Orbany MI. Preoxygenation with tidal volume and deep breathing techniques: the impact of duration of breathing and fresh gas flow. Anesth Analg. 2001 May;92(5):1337-41. doi: 10.1097/00000539-200105000-00049. PMID 11323373